CLINICAL TRIAL: NCT04529447
Title: Hospital Operational Response Strategy and Experience During the COVID-19 Pandemic in a Spine-specialty Korean Medicine Training Hospital
Brief Title: Response of Korean Medicine Hospital to COVID-19
Status: Completed | Type: Observational
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JMA-CT-2020-01
Record Dates: First submitted 2020-08-26; First posted 2020-08-27 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient satisfaction survey: Jaseng Hospital of Korean medicine conducted a pen and paper survey on patient satisfaction with regard to its COVID-19 response in inpatients hospitalized and outpatients visiting during March 23-25, 2020.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The patient satisfaction survey consisted of 8 items, including 7 Likert scale questions and 1 multiple choice question.

SUMMARY:
The objectives of this study are to report the response strategy to prevent COVID-19 spread implemented at a Korean medicine hospital, and the satisfaction survey results regarding its preventive measures.

DETAILED DESCRIPTION:
The objectives of this study are (1) to report the response strategy to prevent COVID-19 spread implemented at a Korean medicine hospital situated in Seoul, Korea, (2) to describe patient visit trends compared to the number of confirmed COVID-19 cases during the COVID-19 peak in February - April 2020, and (3) to provide results of a satisfaction survey regarding its preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients hospitalized at Jaseng Hospital of Korean medicine during March 23-25, 2020
* Outpatients visiting Jaseng Hospital of Korean medicine during March 23-25, 2020

Exclusion Criteria:

* Visitors visiting Jaseng Hospital of Korean medicine during March 23-25, 2020 for purposes other than treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients hospitalized and outpatients visiting Jaseng Hospital of Korean medicine during March 23-25, 2020
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Satisfactory service regarding hospital response to COVID-19 | Baseline (time of current visit)
  Multiple choice question on satisfactory service regarding hospital response to COVID-19, if any

SECONDARY OUTCOMES:
Feelings of apprehension regarding hospital visits | Baseline (time of current visit)
  Likert scale question on level of feelings of apprehension before hospital visits due to COVID-19
Medical staff wearing of facial masks and hand hygiene | Baseline (time of current visit)
  Likert scale question on level of maintenance of wearing of facial masks and hand hygiene in medical staff
Cleanliness and sterilization of hospital facilities | Baseline (time of current visit)
  Likert scale question on level of cleanliness and sterilization of hospital facilities with regard to COVID-19 spread prevention
Convenience and accessibility of hand sanitizers | Baseline (time of current visit)
  Likert scale question on level of convenience and accessibility of hand sanitizers
Helpfulness and readability of posters and stand-up banners | Baseline (time of current visit)
  Likert scale question on level of helpfulness and readability of posters and stand-up banners with COVID-19 information in the hospital
Satisfaction with hospital safety measures for COVID-19 | Baseline (time of current visit)
  Likert scale question on level of satisfaction with hospital safety measures for COVID-19
Recommendation of hospital to friends and family | Baseline (time of current visit)
  Likert scale question on level of recommendation of this hospital to friends and family concerned with visiting hospitals due to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Jinho Lee, KMD, Ph.D., Study Director — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No